CLINICAL TRIAL: NCT05624385
Title: A Feasibility Study of MRgFUS in the Treatment of Therapy-Resistant Tremor-Related Patients With Low SDR Value
Brief Title: MRgFUS Thalamotomy for Therapy-Resistant Tremor-related Disease With Low SDR Value
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRgFUS-Tremor Disorders
Record Dates: First submitted 2022-11-10; First posted 2022-11-22 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Movement Disorders
Keywords: Essential tremor; Parkinson disease; MRgFUS
MeSH Terms: conditions — Movement Disorders; Essential Tremor; Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRgFUS treatment (Experimental)
  Interventions: Device: MRgFUS treatment

INTERVENTIONS:
Device: MRgFUS treatment — ExAblate Transcranial MRgFUS Thalamotomy Treatment of Medication Refractory Tremor-Related Subjects
  Other Names: Thalamotomy

SUMMARY:
A study to evaluate the effectiveness and safety of ExAblate transcranial MRgFUS Thalamotomy treatment of medication refractory tremor-related diseases subjects with low skull density ratio (SDR) value.

Essential tremor (ET) and Parkinson disease (PD) are the most prevalent tremor disorders. ET, considered as a pure tremor disease, is characterized by upper limb intention or postural tremor, while PD is characterized by a variety of motor and non-motor symptoms, among them rest tremor. A number of studies have demonstrated that Magnetic resonance-guided focused ultrasound (MRgFUS) thalamotomy is a minimally invasive and effective procedure suitable for medication-refractory tremor in patients with ET and patients with PD. However, the skull is the main barrier to MRgFUS thalamotomy therapy and patients are screened by calculating SDR value before treatment. The US FDA recommended SDR value >0.45±0.05 as the inclusion criterion for screening patients with tremor treated by MRgFUS system. However, about 20%-50% of patients with SDR value are lower than this standard, which makes this part of patients excluded and unable to accept this treatment with many advantages such as non-invasive, no need for general anesthesia, and no need for hardware implantation. Therefore, this study intended to evaluate the safety and effectiveness of MRgFUS thalamotomy in the treatment of tremor-related patients with low SDR value, so as to provide clinical basis for more patients with tremor to benefit from this treatment.

DETAILED DESCRIPTION:
Patients:

Patients with medication-refractory ET and PD were included. Baseline materials, clinical rating scale for tremor (CRST) , treatment parameters(energy, power, duration time, temperature, target location) , associated adverse effects were recorded.

Imaging protocols:

T2; T2 Flair; DWI; ESWAN; MRS; 3D ASL 2.0s; 3D-T1; DTI; rs-functional MRI Imaging evaluation:

1. Lesion appearance and volume are measured by T2, T2 Flair, DWI, ESWAN, 3D-T1;
2. ESWAN and MRS manifests the changes of iron deposition and metabolism #respectively;
3. ASL shows regional cerebral blood flow associated with the procedure;
4. DTI demonstrates the destruction of white matter integrity.
5. Rs-functional MRI reflects alterations of resting-state brain activity.

Treatment:

MRgFUS thalamotomy

Follow-up:

Baseline (MRI+clinical evaluation); 1-day, 1-month, 3-months, 6-months,1-year, 2-years (MRI+clinical evaluation).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 22 years or older;
2. Subjects are able and willing to agree to participate in the study and can accept all research visits;
3. A diagnosis of ET and PD as confirmed from clinical history and examination by a neurologist or neurosurgeon specialized in movement disorder and intolerance to side effects of medication or poor response to medication, severe and disabling tremor;
4. Able to adapt to MRI system;
5. To tolerate operation with or without some form of sedative (e.g., awake sedation);
6. Able to communicate with the doctor during the operation;
7. Able to use the "Stop ultrasonic processing" button;
8. Skull density ratio (SDR) ≥ 0.28.

Exclusion Criteria:

1. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, known intolerance or allergies to the MRI contrast agent (e.g.Gadolinium or Magnevist) including advanced kidney disease, etc;
2. Pregnant woman;
3. Subjects with severely impaired renal function;
4. Subjects with unstable cardiac status or severe hypertension (diastolic BP > 100 on medication);
5. Subjects show behaviors consistent with alcohol or drug abuse;
6. History of abnormal bleeding and/or coagulopathy/ or intracranial hemorrhage;
7. Patients who received anticoagulant therapy or medications known to increase the risk of bleeding within the month prior to receiving focused ultrasound treatment;
8. Cerebrovascular disease (multiple CVA or CVA within 3 months);
9. Subjects with brain tumors.
10. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (can be up to 2 hrs of total time).

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
1.1 Safety To evaluate the incidence and severity of adverse events (AE/AEs) associated with ExAblate Transcranial MRgFUS treatment of subjects during 2-year follow-up. | 2 years
  All AE reported by the investigator are classified as: definitely relevant, very likely relevant, probably relevant, probably not relevant or definitely not relevant to the product under study, where definitely relevant, very likely relevant, possibly relevant are classified as relevant, probably not relevant and definitely not relevant are classified as irrelevant.

SECONDARY OUTCOMES:
2.1. Safety To evaluate the incidence and severity of adverse events (AE/AEs) after ExAblate Transcranial MRgFUS treatment of subjects at 24 hours, 1 month, 3 months, 6 months, 12 months, and 2 years follow-up. | 2 years
  To evaluate the incidence of unexpected adverse device events (UADE) within 2 years after the treatment of the study product.
2.2. Effectiveness | 2 years
  The effectiveness will be evaluated by the hand tremor subscore (on a scale ranging from 0 to 32 when the dominant hand is treated and 0 to 28 points when the nondominant hand is treated, with higher scores indicating more severe tremor), which was derived from the Clinical Rating Scale for Tremor (CRST) . Both the treatment side and the non-treatment side of the subject will be evaluated.
  Clinical evaluation will be conducted at the following time points: at screening, at baseline, and 1, 3, 6, 12 months, and 2 years after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China